CLINICAL TRIAL: NCT04976660
Title: Phase I/II First-in-Human Study of TT-4 As a Single Agent in Participants with Advanced Selected Solid Tumors
Brief Title: TT-4 As a Single Agent in Subjects with Advanced Selected Solid Tumors
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Tarus is conducting clinical development under a single IND, specifically IND for TT-10 (PORT-6). Tarus has withdrawn Study TT-4-101 under the TT-4 IND; however the TT-4 IND will remain active.
Sponsor: Tarus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Organization: Portage Biotech (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TT-4-101
Record Dates: First submitted 2021-07-06; First posted 2021-07-26 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer; Gastric Cancer; Hepatocellular Carcinoma; Pancreatic Cancer
Keywords: failed or not eligible for standard of care; Advanced Selected Solid Tumors; TT-4; Adenosine; Adenosine Antagonist; A2B; A2BR Inhibitor
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Carcinoma, Hepatocellular; Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: 3+3 Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multiple Ascending Dose (Experimental): 3+3 Dose escalation until MTD and/or R2PD of TT-4 is determined
  Interventions: Drug: TT-4

INTERVENTIONS:
Drug: TT-4 — TT-4 orally administered QD starting at 200 mg and will be increased to 800 mg (dosing may be increased to BID, if appropriate based on emerging safety, PK or PD data).

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of orally administered TT-4 in subjects with advanced selected solid tumors. The dose escalation portion of the study will determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of TT-4.

DETAILED DESCRIPTION:
Multicenter, open-label dose-escalation Phase I/II clinical study, designed to evaluate the safety, tolerability, PK, PD, anti-tumor activity, and efficacy of TT-4 in subjects diagnosed with Colorectal Cancer (CRC), Gastric cancer (GC), Hepatocellular Carcinoma (HCC) and locally advanced, unresectable, or metastatic Pancreatic Cancer (PANC); who have failed or are not eligible for standard of care treatment.

The study will be conducted in two phases. Dose escalation (Phase 1) will be to determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D), safety and tolerability of TT-4 in subjects with advanced subjects diagnosed with Colorectal Cancer (CRC), Gastric cancer (GC), Hepatocellular Carcinoma (HCC) and locally advanced, unresectable, or metastatic Pancreatic Cancer (PANC); who have failed or are not eligible for standard of care treatment. Dose expansion (Phase 2) will be to further explore the safety and tolerability of the MTD and/or RP2D, PK, PD, antitumor activity, and efficacy of TT-4.

ELIGIBILITY:
Inclusion Criteria

To eligible for inclusion in the dose escalation cohort or expansion cohort 1 in this study, subjects must meet all of the following criteria:

1. Subjects must be ≥18 years of age.
2. Subjects or their legal representative must be able to provide written informed consent to participate in the trial prior to the performance of any study-specific procedures.
3. Diagnosis of histologically or cytologically confirmed advanced selected solid tumors

   * Cohort A dose escalation: Colorectal Cancer, Gastric cancer, Hepatocellular Carcinoma and locally advanced, unresectable, or metastatic Pancreatic Cancer, who have failed or are not eligible for standard of care treatment.
   * Cohort B: Advanced colorectal cancer (CRC), who have failed or not eligible for standard of care
   * Cohort C: Advanced Gastric cancer (GC), who have failed or not eligible for standard of care
   * Cohort D: Advanced Hepatocellular Carcinoma (HCC), who have failed or not eligible for standard of care
   * Cohort E: Locally advanced, unresectable, or metastatic Pancreatic Cancer (PANC), who have failed or not eligible for standard of care
4. ECOG performance status (PS) score 0-1
5. Have measurable disease per RECIST 1.1 or (for subjects in the expansion cohorts) iRECIST as assessed by the local site investigator/radiology. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
6. Subjects must have locally advanced, recurrent or metastatic neoplastic disease that is not curable by currently available therapies.
7. Failure to respond to standard therapy, or for whom no appropriate therapies are available (based on the judgment of the Investigator)
8. Life expectancy of ≥ 3 months
9. Subjects must have adequate hematologic function based on the following:

   * Absolute neutrophil count ≥ 1.5 x 109/L
   * Platelet count ≥ 100 x 109/L
   * Hemoglobin ≥ 9.0 g/dL
10. Subjects must have adequate hepatic function based on the following:

    * Total bilirubin <1.5 × upper limit of normal (ULN) Patients with a known history of Gilbert's syndrome (≤ 3.0 × ULN) and/or isolated elevations of indirect bilirubin are eligible for study participation
    * Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤2.5 x ULN (≤5 × ULN for subjects with known hepatic metastases)
11. Subjects must have adequate renal function based on the following:

    - Serum creatinine ≤1.5 × ULN
12. For women of childbearing potential (WCBP): negative serum β human chorionic gonadotropin (βhCG) pregnancy test within 1 week before first treatment (WCBP defined as a sexually mature woman who has not undergone surgical sterilization or who has not been naturally post-menopausal for at least 12 consecutive months for women > 55 years of age)
13. Human immunodeficiency virus (HIV) infected subjects must be on antiretroviral therapy (ART) and have a well-controlled HIV infection/disease defined as:

    1. Subjects on ART must have a CD4+ T cell count >350 cells/mm3 at time of screening
    2. Subjects on ART must have achieved and maintained virologic suppression defined as confirmed HIV RNA level below 50 copies/mL or the lower limit of qualification (below the limit of detection) using the locally available assay at the time of screening and for at least 12 weeks prior to screening
    3. Subjects on ART must have been on a stable regimen, without changes in drugs or dose modification, for at least 4 weeks prior to study entry (Day 1).
14. For women of childbearing potential (WCBP): negative urine pregnancy test (UPT) within 1 week before first treatment (WCBP defined as a sexually mature woman who has not undergone surgical sterilization or who has not been naturally post-menopausal for at least 12 consecutive months for women > 55 years of age). WCBP should be placed on effective birth control directly after testing negative for pregnancy; if not, then WCBP should have a UPT on Day 1 of every cycle, prior to drug administration. Any positive or indeterminant UPT result must be confirmed by Serum.
15. Female subjects of childbearing potential must use a highly effective mode of contraception or abstain from heterosexual activity for the duration of the trial and for 120 days following the last dose of study medication. A female is NOT of childbearing potential if she has undergone bilateral salpingoophorectomy or is menopausal, defined as an absence of menses for 12 consecutive months. Male subjects must agree to use highly effective contraception.
16. Ability to adhere to the study visit schedule and all protocol requirements

Exclusion Criteria

Subjects are to be excluded from the study if they meet any of the following criteria:

1. Major surgery within 4 weeks prior to Screening
2. Anti-cancer therapy, such as chemotherapy, immunotherapy, hormonal therapy, targeted therapy, or investigational agents within five half-lives or four weeks, whichever is shorter, prior to administration of the first dose of study treatment.
3. Subjects with active central nervous system (CNS) metastases; however, subjects who have undergone radiation and/or surgery for the treatment of CNS metastases, who are neurologically stable, and who are no longer taking pharmacologic doses of corticosteroids are eligible; subjects with leptomeningeal metastases are not eligible.
4. Has received prior radiotherapy within 2 weeks of start of study treatment. Subjects must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
5. Primary CNS malignancy
6. HIV-infected subjects with a history of Kaposi sarcoma and/or Multicentric Castleman Disease.
7. Subjects who are hepatitis B surface antigen positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to enrollment.

   Note: Subjects should remain on antiviral therapy throughout study intervention and follow local guidelines for HBV antiviral therapy post completion of study intervention.

   Hepatitis B screening tests are not required unless:
   * Known history of HBV infection
   * As mandated by local health authority.
8. Subjects with a history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening. Note: Subjects must have completed curative antiviral therapy at least 4 weeks prior to enrollment.

   Hepatitis C screening tests are not required unless:
   * Known history of HCV infection
   * As mandated by local health authority.
9. Subjects who require immunosuppressive therapy including, but not limited to, treatment with corticosteroids in pharmacologic doses (equivalent to ≥10 mg prednisone daily), cyclosporine, mycophenolate, azathioprine, methotrexate, adalimumab, infliximab, vedolizumab, tofacitinib, dupilumab, rituximab, etc. or systemic steroids (except for steroid use as cortisol replacement therapy in documented adrenal insufficiency)
10. Ongoing systemic bacterial, fungal, or viral infections at Screening

    a. NOTE: Subjects on antimicrobial, antifungal, or antiviral prophylaxis are not specifically excluded if all other inclusion/exclusion criteria are met
11. Administration of a live vaccine within 30 days of first dose of study drug
12. Baseline QT interval corrected with Fridericia's method (QTcF) > 480 ms (average of triplicate readings)

    a. NOTE: Criterion does not apply to subjects with a right or left bundle branch block.
13. Subjects with a history of Torsade de Pointes or taking QT-prolonging drugs
14. Prior surgery or gastrointestinal dysfunction that may affect drug absorption (eg, gastric bypass surgery, gastrectomy)
15. Female subjects who are pregnant or breastfeeding
16. Concurrent active malignancy other than non-melanoma skin cancer, carcinoma in situ of the cervix, or prostate intraepithelial neoplasia
17. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease
18. History of peptic ulcer and/or gastrointestinal bleed within the past 6 months prior to Screening
19. History of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the last 6 months prior to Screening
20. Unstable or severe uncontrolled medical condition (eg, unstable cardiac function, unstable pulmonary condition including pneumonitis and/or interstitial lung disease, uncontrolled diabetes) or any important medical illness or abnormal laboratory finding that would, in the Investigator's judgment, increase the risk to the subject associated with his or her participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with Dose Limiting Toxicities (DLTs) of TT-4 during the dose escalation phase | 28 Days
  All toxicities will be graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Define the maximum tolerated dose (MTD) or phase 2 recommended dose of TT-4during the dose escalation phase | Up to 1 year
Overall Response Rate (ORR) | From study enrollment until participant discontinuation, first occurrence of progressive disease, or death from any cause, whichever occurs first (approximately 2 years)
  This is defined as complete response (CR) or PR according to RECIST 1.1 and from the first dose until documented confirmed disease progression.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) overall and by severity, seriousness and relatedness. | Through study completion, an average of 1 year
  Safety assessments will be performed on a regular basis using physical examination, spontaneous AE reporting, scheduled and unscheduled laboratory assessments, and other diagnostic evaluations as indicated. Adverse events will be reported using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Duration of Response (DoR) | From study enrollment until participant discontinuation, first occurrence of progressive disease, or death from any cause, whichever occurs first (approximately 2 years)]
  Time from first confirmed documented objective response (CR or PR) to the date of first confirmed documented objective progression of disease (PD) or death due to any cause whichever occurs first. If a subject has not had an event (PD or death), DR is censored at the date of last adequate tumor assessment.
Progression Free Survival (PFS) | From study enrollment until participant discontinuation, first occurrence of progressive disease, or death from any cause, whichever occurs first (approximately 2 years)]
  Time from first dose to the date of the first confirmed documented objective progression of disease (PD) or death due to any cause, whichever occurs first.
Peak serum concentration (Cmax) of TT-4 | Predose, 0.5, 1, 2, 4, 6, 8, 24 hours post-dose
  PK Parameter
Area under the serum concentration versus time curve (AUC) of TT-4 | Predose, 0.5, 1, 2, 4, 6, 8, 24 hours post-dose
  PK Parameter
Half-life of TT-4 | Predose, 0.5, 1, 2, 4, 6, 8, 24 hours post-dose
  PK Parameter

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Antonioli L, Blandizzi C, Pacher P, Hasko G. Immunity, inflammation and cancer: a leading role for adenosine. Nat Rev Cancer. 2013 Dec;13(12):842-57. doi: 10.1038/nrc3613. Epub 2013 Nov 14. PMID 24226193
- [Background] Cekic C, Sag D, Li Y, Theodorescu D, Strieter RM, Linden J. Adenosine A2B receptor blockade slows growth of bladder and breast tumors. J Immunol. 2012 Jan 1;188(1):198-205. doi: 10.4049/jimmunol.1101845. Epub 2011 Nov 23. PMID 22116822
- [Background] Aherne CM, Kewley EM, Eltzschig HK. The resurgence of A2B adenosine receptor signaling. Biochim Biophys Acta. 2011 May;1808(5):1329-39. doi: 10.1016/j.bbamem.2010.05.016. Epub 2010 May 28. PMID 20546702
- [Background] Allard B, Allard D, Buisseret L, Stagg J. The adenosine pathway in immuno-oncology. Nat Rev Clin Oncol. 2020 Oct;17(10):611-629. doi: 10.1038/s41571-020-0382-2. Epub 2020 Jun 8. PMID 32514148
- [Background] Zhou Y, Chu X, Deng F, Tong L, Tong G, Yi Y, Liu J, Tang J, Tang Y, Xia Y, Dai Y. The adenosine A2b receptor promotes tumor progression of bladder urothelial carcinoma by enhancing MAPK signaling pathway. Oncotarget. 2017 Jul 25;8(30):48755-48768. doi: 10.18632/oncotarget.17835. PMID 28548944
- [Background] Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, Lin NU, Litiere S, Dancey J, Chen A, Hodi FS, Therasse P, Hoekstra OS, Shankar LK, Wolchok JD, Ballinger M, Caramella C, de Vries EGE; RECIST working group. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol. 2017 Mar;18(3):e143-e152. doi: 10.1016/S1470-2045(17)30074-8. Epub 2017 Mar 2. PMID 28271869
- [Background] Horigome E, Fujieda M, Handa T, Katayama A, Ito M, Ichihara A, Tanaka D, Gombodorj N, Yoshiyama S, Yamane A, Yamada K, Horiguchi J, Shinozuka K, Oyama T, Nishiyama M, Rokudai S. Mutant TP53 modulates metastasis of triple negative breast cancer through adenosine A2b receptor signaling. Oncotarget. 2018 Oct 2;9(77):34554-34566. doi: 10.18632/oncotarget.26177. eCollection 2018 Oct 2. PMID 30349649
- [Background] Vecchio EA, Tan CY, Gregory KJ, Christopoulos A, White PJ, May LT. Ligand-Independent Adenosine A2B Receptor Constitutive Activity as a Promoter of Prostate Cancer Cell Proliferation. J Pharmacol Exp Ther. 2016 Apr;357(1):36-44. doi: 10.1124/jpet.115.230003. Epub 2016 Jan 20. PMID 26791603
- [Background] Lan J, Lu H, Samanta D, Salman S, Lu Y, Semenza GL. Hypoxia-inducible factor 1-dependent expression of adenosine receptor 2B promotes breast cancer stem cell enrichment. Proc Natl Acad Sci U S A. 2018 Oct 9;115(41):E9640-E9648. doi: 10.1073/pnas.1809695115. Epub 2018 Sep 21. PMID 30242135
- [Background] Ma DF, Kondo T, Nakazawa T, Niu DF, Mochizuki K, Kawasaki T, Yamane T, Katoh R. Hypoxia-inducible adenosine A2B receptor modulates proliferation of colon carcinoma cells. Hum Pathol. 2010 Nov;41(11):1550-7. doi: 10.1016/j.humpath.2010.04.008. PMID 20619442
- [Background] Ryzhov S, Novitskiy SV, Zaynagetdinov R, Goldstein AE, Carbone DP, Biaggioni I, Dikov MM, Feoktistov I. Host A(2B) adenosine receptors promote carcinoma growth. Neoplasia. 2008 Sep;10(9):987-95. doi: 10.1593/neo.08478. PMID 18714400